CLINICAL TRIAL: NCT03091452
Title: CArdioSurgEry Atrial Fibrillation Register - CASE-AF Register
Brief Title: CArdioSurgEry Atrial Fibrillation Register
Acronym: CASE-AF
Status: Recruiting | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: CASE-AF
Record Dates: First submitted 2017-03-13; First posted 2017-03-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CASE AF aims to describe the reality of medical care of patients in whom atrial fibrillation is treated by cardiac surgical ablation.

DETAILED DESCRIPTION:
CASE AF aims to describe the reality of medical care of patients in whom atrial fibrillation is treated by cardiac surgical ablation. In particular, the following questions should be answered:

* Indication: Which are the different indications for cardiac surgical ablation in patients with atrial fibrillation?
* How often and in which patients the different concepts of surgery and ablation procedures are used? At the same time, how often an intervention at the left atrial appendage is carried out?
* Safety: How secure is the cardiac surgical ablation of atrial fibrillation (periprocedural, during hospital stay and during the long-term follow up)?
* Effectiveness: How effectively is the cardiac surgical ablation of atrial fibrillation (procedural success)? How often are AF recurrences in the long-term follow up?
* What is the concommitant medical treatment after surgical ablation?

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrilation
* Treated by cardiac surgical ablation

Exclusion Criteria:

* Patient denies participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom atrial fibrillation is treated by cardiac surgical ablation
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of major bleeding events | 12 months
  Documentation of procedural results and clinical short-and long-term results of the documented therapies

SECONDARY OUTCOMES:
Number of major adverse cardiac events | 12 months
  Documentation of procedural results and clinical short-and long-term results of the documented therapies
Complications during hospital stay | 12 months
  Documentation of hospital mortality, nonfatal major complications

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Hanke, MD, Principal Investigator — Asklepios Hamburg Harburg
Locations (3):
- Germany (3):
  - Klinikum Bogenhausen, München, Bavaria
  - Asklepios Harburg, Hamburg, Hamburg
  - Schüchtermann Kliniken, Bad Rothenfelde, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No